CLINICAL TRIAL: NCT03341533
Title: Abdominal Ice Packs for Pain Control and Reduction of Narcotic Use Following Laparoscopic Hysterectomy: A Randomized Controlled Trial
Brief Title: Abdominal Ice Packs for Pain Control and Reduction of Narcotic Use Following Laparoscopic Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Tatnai L. Burnett, Senior Associate Consultant, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-007182
Record Dates: First submitted 2017-11-08; First posted 2017-11-14 (Actual); Results first posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Pain, Postoperative; Hysterectomy; Narcotic Use; Cryotherapy Effect
Keywords: Analgesia; Laparoscopy; Pain
MeSH Terms: conditions — Pain, Postoperative; Agnosia; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ice packs plus usual post-op analgesia (Experimental): Ice pack applied to the abdomen and maintained continuously for the first 12 hours post-operatively. Standard standard post-operative analgesia orders will be followed in addition to use of ice.
  Interventions: Procedure: Ice packs plus usual post-op analgesia; Other: Usual post-op analgesia
- Usual post-op analgesia (Active Comparator): Standard post-operative analgesia only, no ice use.
  Interventions: Other: Usual post-op analgesia

INTERVENTIONS:
Procedure: Ice packs plus usual post-op analgesia — A 9 inch by 12 inch zip lock bag filled with ice chips, placed inside a cotton pillow case, placed directly on the abdomen. Ice chips will be replaced as they thaw. Monitoring of surgical sites, skin integrity, and comfort with ice pack in place by nursing per current procedural guidelines.
  Arms: Ice packs plus usual post-op analgesia
Other: Usual post-op analgesia — Standard post-operative analgesia orders will be followed.

SUMMARY:
The purpose of this study is to evaluate the effect of using ice packs on the abdomen immediately after laparoscopic hysterectomy surgery on pain control and narcotic pain medication use.

DETAILED DESCRIPTION:
Hysterectomy is one of the most common surgical procedures performed on women in the United States, with approximately 600,000 performed annually. The use of postoperative cooling as an adjuvant for post-operative pain control has previously been shown to be effective and safe in a variety of procedures, but has yet to be described for laparoscopic surgery. In contrast to laparotomy where the wound is a significant pain generator and direct application of ice is intuitive, in laparoscopic surgery much of the pain-generating tissue trauma is intraperitoneal and pelvic in nature, away from the abdominal wall. Ice pack use on the abdominal wall likely inhibits visceral afferent pain fibers via somatic afferent nerve cross-talk. Accordingly, applying ice to the abdominal wall and its somatic afferents may improve laparoscopic pain control, despite the lack of a significant abdominal wound. Our goal is to quantify narcotic use after hospital discharge following hysterectomy, and evaluate the effectiveness of abdominal ice packs as low cost adjuncts for pain control.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing robotic or conventional laparoscopic hysterectomy

Exclusion Criteria:

* Any opioid use within 2 weeks of surgery date
* Planned post-operative ICU admission
* Conversion of laparoscopic approach to laparotomy or any incision ≥4 cm
* Regional anesthesia/analgesia, including tap block use

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2019-04-05 (Actual); Study Completion 2020-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tatnai L. Burnett, M.D., Principal Investigator — Obstetrics and Gynecology
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cope AG, Wetzstein MM, Mara KC, Laughlin-Tommaso SK, Warner NS, Burnett TL. Abdominal Ice after Laparoscopic Hysterectomy: A Randomized Controlled Trial. J Minim Invasive Gynecol. 2021 Feb;28(2):342-350.e2. doi: 10.1016/j.jmig.2020.06.027. Epub 2020 Jul 3. PMID 32622918
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ice Packs Plus Usual Post-op Analgesia | Usual Post-op Analgesia
Started | 72 | 70
Completed | 69 | 68
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Not eligible after randomization | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ice Packs Plus Usual Post-op Analgesia | Usual Post-op Analgesia | Total
Number analyzed (Participants) | 69 | 68 | 137
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (11.1) | 56.9 (13) | 57.1 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 68 | 137
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 68 | 66 | 134
  Other | 1 | 0 | 1
  Choose Not to Disclose | 0 | 1 | 1
  Unknown | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 69 | 68 | 137

OUTCOME MEASURES:

1. Primary Outcome: Numeric Pain Intensity Scale
Description: Self-reported pain intensity scores (Numerical Pain Intensity Scale, 0-10 visual analog scale with 0 representing no pain and 10 representing the worst pain imaginable) assessed and documented a minimum every four hours post-operatively. Mean differences of pain intensity assessed between ice group and usual care group.
Time Frame: 12 hours post-operatively
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ice Packs Plus Usual Post-op Analgesia | Usual Post-op Analgesia
Number analyzed (Participants) | 69 | 68
score on a scale | 3 [1 to 4] | 3 [2 to 4]
Statistical Analysis 1: Comparison: Ice Packs Plus Usual Post-op Analgesia vs Usual Post-op Analgesia; Test type: Equivalence — The null hypothesis is that there is no difference in NPIS between the two groups; p = 0.39, Kruskal-Wallis; difference in medians = 0.0

2. Primary Outcome: Mean Morphine Metabolic Equivalents (MME) Consumption: Inpatient Floor
Description: Calculation of average patient MME from the time enter hospital floor to hospital discharge. Administered narcotics will be abstracted from the medical record and converted to total MME for analysis.
Time Frame: an average of one day from entering hospital floor to discharge
Measure: Median (Full Range); unit: MME
Arm/Group | Ice Packs Plus Usual Post-op Analgesia | Usual Post-op Analgesia
Number analyzed (Participants) | 69 | 68
MME | 7.5 [0 to 67.5] | 12 [0 to 67.5]
Statistical Analysis 1: Comparison: Ice Packs Plus Usual Post-op Analgesia vs Usual Post-op Analgesia; Test type: Equivalence — The null hypothesis is that there is no difference in MME use on the hospital floor between groups; p = 0.88, Kruskal-Wallis; Difference of medians = -4.5 — Ice packs - Usual care

3. Secondary Outcome: Mean Morphine Metabolic Equivalents (MME) Consumption: Outpatient
Description: Calculation of average patient MME from the time of hospital discharge to end of narcotic use for post-operative pain control. Patients will keep detailed home diary of narcotic analgesia use after discharge. Total narcotic intake recorded on the diary will be converted to MME for analysis.
Time Frame: 2 weeks
Population: Some patients (N=6 ice pack patients and N=6 usual care patients) kept a diary of at home narcotic use after discharge as directed, which is why the numbers for this analysis are lower than the total number of patients.
Measure: Median (Full Range); unit: MME
Arm/Group | Ice Packs Plus Usual Post-op Analgesia | Usual Post-op Analgesia
Number analyzed (Participants) | 63 | 62
MME | 29.5 [0 to 224.9] | 26.5 [0 to 175]
Statistical Analysis 1: Comparison: Ice Packs Plus Usual Post-op Analgesia vs Usual Post-op Analgesia; Test type: Equivalence — The null hypothesis is that the outpatient MME consumption will be the same across the two groups; p = 0.75, Kruskal-Wallis; difference in medians = -7.5 — Ice packs - Usual Care

4. Secondary Outcome: Brief Pain Inventory Short Form - Postoperative Pain Severity
Description: Brief Pain Inventory Short Form scores (Pain diagram to indicate location of pain and 7 Likert-scale questions assessing pain severity and interference with feeling and function, scores ranging from 0 = No pain to 10 = pain as bad as you can imagine) assessed pre-op and again post-operatively, just before hospital discharge (at last 12 but no more than 24 hours after surgery). Mean differences calculated between ice group and usual care group.
Time Frame: one day after surgery
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ice Packs Plus Usual Post-op Analgesia | Usual Post-op Analgesia
Number analyzed (Participants) | 67 | 68
score on a scale | 3 [2 to 4] | 3.3 [2.1 to 4.3]
Statistical Analysis 1: Comparison: Ice Packs Plus Usual Post-op Analgesia vs Usual Post-op Analgesia; Test type: Equivalence — The null hypothesis is that the postoperative BPI pain severity score will be the same between groups; p = 0.80, Kruskal-Wallis; difference in medians = -0.3 — Ice Packs - Usual Care

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from immediately after the operation until the scheduled 6 - 8 week postoperative visit. Systematic assessment for occurrence of adverse events was performed by study personnel at all points of contact during the postoperative course and by record review.
Arm/Group | Ice Packs Plus Usual Post-op Analgesia | Usual Post-op Analgesia
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/70
Serious Adverse Events (participants affected / at risk) | 3/72 | 4/70
Other Adverse Events (participants affected / at risk) | 5/72 | 5/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ice Packs Plus Usual Post-op Analgesia (N=72) | Usual Post-op Analgesia (N=70)
Vaginal cuff dehiscence (Surgical and medical procedures) | 1 (1) | 1 (1)
Vaginal cuff bleeding (Surgical and medical procedures) | 0 (0) | 2 (2)
Postoperative Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bowel injury and subsequent sepsis (Surgical and medical procedures) | 1 (1) | 0 (0)
Wound infection (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ice Packs Plus Usual Post-op Analgesia (N=72) | Usual Post-op Analgesia (N=70)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 1 (1)
Nause (Gastrointestinal disorders) | 0 (0) | 1 (1)
New onset pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Skin erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Related to ice
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Postoperative fever and pain (Surgical and medical procedures) | 1 (1) | 0 (0)
Allergic reaction to medication (Immune system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT03341533/Prot_SAP_ICF_000.pdf